CLINICAL TRIAL: NCT06101602
Title: Immediate Effect of Dynamic Stretching With and Without Floss Band on Flexibility of Hamstrings in Futsal Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/01382 Shiza Fatima Zaidi
Record Dates: First submitted 2023-10-11; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Sports Physical Therapy
Keywords: Dynamic Stretching; Flexibility; Flossing; Hamstring Muscles; Soccer; Sports Injuries
MeSH Terms: conditions — Athletic Injuries | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Concurrent Parallel Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With Floss Band (Experimental): Floss band made of natural rubber, black in color and 4" in width will be wrapped around the thigh, starting from the distally to superiorly with an overlap of 50%. Perform exercises:
  • Multi-directional leg swing
  Interventions: Other: Dynamic Stretching with Floss Band
- Without floss Band (Active Comparator): Perform exercises without floss band.
  • Multi-directional leg swing
  Interventions: Other: Dynamic Stretching without Floss Band

INTERVENTIONS:
Other: Dynamic Stretching with Floss Band — Floss band involves wrapping a band made of natural rubber around the targeted joint or muscle for 1-3 minutes through active movement. The mechanism behind flossing is thought to have a "three-fold effect", compression may stimulate the mechanoreceptors of the underlying fascia layer which causes the hyperemia of the targeted tissue, and leads to increased blood flow.
  This intervention was applied in addition to dynamic stretching which involved 3 types of dynamic stretches. These stretches were applied through multidirectional (anteromedial, anterior, and anterolateral) leg swings specifically for the Hamstring muscle. It was performed in 3 sets of 15 repetitions with 30 seconds of rest between each exercise.
  Arms: With Floss Band
Other: Dynamic Stretching without Floss Band — In this group, only dynamic stretching was applied which involved 3 types of dynamic stretches. These stretches were applied through multidirectional (anteromedial, anterior, and anterolateral) leg swings specifically for the Hamstring muscle. It was performed in 3 sets of 15 repetitions with 30 seconds of rest between each exercise.
  Arms: Without floss Band

SUMMARY:
To compare the immediate effect of dynamic stretching with and without floss band on the hamstring flexibility in futsal players.

DETAILED DESCRIPTION:
Futsal is a soccer-like indoor sport that has been gaining popularity worldwide.To increase the flexibility and ROM of involved muscle group a new method has been introduced named Flossing of tissue by using a floss band.

This research study will be helpful to enable therapists to broaden their treatment plans or choose better treatment tools for improving hamstrings flexibility in futsal players. Thus, this study has been designed with the purpose to examine the effect of dynamic stretching with and without floss band on the flexibility of the hamstring.

ELIGIBILITY:
Inclusion Criteria:

* National level futsal players.
* Active for past 3 months.

Exclusion Criteria:

* Players with any systemic disease/disorder.
* Players with any recent ligamentous or musculoskeletal injury that isn't healed yet.

Ages: 17 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Straight Leg Raise (SLR) Test | Baseline and immediately after the intervention
  Universal goniometer was used to measure SLR angle.
Active Knee Extension (AKE) Test | Baseline and immediately after the intervention
  Universal goniometer was used to measure AKE angle.
Sit and Reach Test | Baseline and immediately after the intervention
  A ruler was used to measure Sit and Reach Test Score.

SECONDARY OUTCOMES:
Serum Creatine Kinase (CK) Levels | Baseline and after 24 hours of the intervention
  Creatine-kinase is a type of enzyme that muscle cell need to function, small amount of CK is present in our blood but high level indicates muscle injury. CK-MM is the substance rises when skeletal muscle is injured. This test is valid(r=0.58) and reliable (r=0.87) to check the muscle damage.
Serum Lactate Dehydrogenase (LDH) levels | Baseline and after 24 hours of the intervention
  Lactate Dehydrogenase is an enzyme found in body and it converts sugar into energy. When a tissue is damaged, the level of this enzyme in blood increases. This test is valid (r=0.98) to check the muscle damage

CONTACTS AND LOCATIONS:
Overall Officials: Noman Sadiq, MS-SPT, Principal Investigator — Riphah International University, Islamabad.
Locations (1):
- Riphah International University (RIU), Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No